CLINICAL TRIAL: NCT06513247
Title: Feasibility of a Pilot Screening Program for Type 1 Diabetes in a High-Risk Population
Brief Title: Screening Program for Type 1 Diabetes in a High-Risk Population
Status: Recruiting | Type: Observational
Sponsor: King Saud University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Reem Al Khalifah, Associate Professor, King Saud University
Other Study IDs: NICS-2024-04-04
Record Dates: First submitted 2024-07-07; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes
Keywords: screening; early detection; ADAP
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — HLA phenotyping and genetic risk score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: screening for Islet autoantibody — IAA, GADA, IA-2A, Zn-transporter 8 autoantibodies
Diagnostic Test: HLA phenotype and genetic risk score — using DBS filter paper

SUMMARY:
Type 1 diabetes mellitus (T1D) is a growing public health concern in Saudi Arabia, ranking ninth globally in T1D incidence and tenth in T1D prevalence in children, and the rates are expected to rise and incur greater healthcare costs. Genetic and immunological factors are believed to play a significant role in disease development, and recent clinical trials have shown promise in delaying or preventing T1D onset in high-risk individuals. Early screening for immunological or genetic markers in children is crucial to identify high-risk individuals and provide early intervention. Last year, the American diabetes association's recommended clinicians to screen first degree relatives of individual with T1D. Unfortunately, Saudi Arabia and other Arab countries lack established T1D screening programs, making early identification and intervention challenging. The benefits of screening include education for symptom awareness, monitoring to track progression to clinical T1D, a five-fold reduction in diabetic ketoacidosis (DKA) at onset, and improved glucose control for the first years following diagnosis. To address this issue, exploring effective and efficient screening methods in identifying high-risk children and the cultural acceptability, feasibility, and barriers to a broader implementation of such screening programs among Saudi families is crucial. Therefore, the investigators aim to conduct a prospective cohort study among young children and adolescents with a family history of T1D (i.e., T1D first-degree relatives). Children 2-18 years old will be screened using a 5 spots filter-dried blood sample for the following:

1. Islet autoantibodies: IAA, GADA, IA-2A, Zn-transporter autoantibodies using the antibody detection by agglutination PCR (ADAP) assay.
2. HLA phenotyping
3. Genetic risk score after the cross-sectional assessment those who are determined to be in stage I, or II of T1D will be offered prospective follow-up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis in a first-degree relative:

Diabetes is defined based on the American diabetes association (ADA) definition: Classic symptoms of diabetes or hyperglycemic crisis, with plasma glucose concentration ≥11.1 mmol/L (200 mg/dL), or Fasting plasma glucose ≥7.0 mmol/L (≥126 mg/dL). Fasting is defined as no caloric intake for at least 8 h, or Two-hour post load glucose ≥11.1 mmol/L (≥200 mg/dL) during an OGTT, or HbA1c >6.5%.

Exclusion Criteria:

* first-degree relative case with Maturity-Onset Diabetes of the Young (MODY) or Type 2 Diabetes Mellitus (T2DM).
* Non-Saudi children.
* first-degree relative not following at our centre.

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 2-18 years old health children with first-degree relatives with T1D.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2024-05-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of stage I, II and III T1D in screened participants. | 6 months
Rates of screening refusal. | 6 months
  measured as number of participants that they refused to be screened.

SECONDARY OUTCOMES:
Rate of completed screened cases | 12 months
  measured as number of participants who complete the screening.
Adverse events associated with the screening process | 6 months
Estimated costs for T1D screening per participant. | 5 years
Estimated costs for DKA | 5 years
Parental anxiety from T1D screening | 1 year
  measured by the generalized anxiety disorder -7 scale (GAD-7)
Glycemic changes among positively screened participants | 5 years
  measured by oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- The University Diabetes Centre at King Saud University Medial CIty, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The data is available from the PI upon reasonable request and approval by the IRB.

REFERENCES:
- [Derived] Algadi IS, AlRuthia Y, Mujammami MH, Aburisheh KH, Alotaibi M, Al Issa S, Al-Saif AA, Seftel D, Tsai CT, Al Khalifah RA. Early Detection of Type 1 Diabetes in First-Degree Relatives in Saudi Arabia (VISION-T1D): Protocol for a Pilot Implementation Study. JMIR Res Protoc. 2025 Apr 14;14:e70575. doi: 10.2196/70575. PMID 39930327